CLINICAL TRIAL: NCT02760966
Title: Effectiveness of Alcohol 70º Compared With Soap on Cord Separation Time and the Complication Rate in the Newborn
Brief Title: Effectiveness of Alcohol 70º vs Soap on Cord Separation Time and the Complication in the Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-ALC-2015-27
Record Dates: First submitted 2016-04-01; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Umbilical Cord
MeSH Terms: interventions — Ethanol; Soaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol 70º (Experimental): Umbilical cord care will be carried out using alcohol 70º at least 3 times a day. Firstly, there must be a proper hand hygiene. Then, with sterile gauzes alcohol will be applied from the abdominal part to the end of the stump.
  Interventions: Other: Alcohol 70º
- Soap (Active Comparator): Umbilical cord care will be carried out using soap at least 3 times a day. Firstly, there must be a proper hand hygiene. Then, with sterile gauzes alcohol will be applied from the abdominal part to the end of the stump.
  Interventions: Other: Soap

INTERVENTIONS:
Other: Alcohol 70º
  Arms: Alcohol 70º
Other: Soap
  Other Names: Jabón neutro
  Arms: Soap

SUMMARY:
Evaluate the effectiveness of alcohol 70º compared with soap on cord separation time and the complication rate in the newborn.

DETAILED DESCRIPTION:
Randomized clinical trial, which objective is to assess the effectiveness of 70º alcohol compared with neutral soap on the cord separation time of a selection of newborns. 34 newborns admitted to the maternity ward of the hospital have participated. The study is divided into two phases, hospital and home. The first stage is located in the hospital, where the patients who will become part of the study are chosen. After receiving the informed letting of the legal guardian the second part of this phase is started; which aim is to explain the steps to be followed to make a correct cleaning cord technique. The home phase consists of being in contact with the family through Whatsapp on the 5th day from birth, the day of the cord fall and 5 days after this fall. Making some simple questions with simple answers such as yes or no and with the possibility, or not, of sending a picture of the cord state in each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Availability of legal guardians with knowledge and access to Whatsapp.

Exclusion Criteria:

* Admission in the newborn's room.
* Patients with strong concomitant illness, that limits the planned activities or whose current state contraindicates the incorporation of the program.
* Mother's age < 18 years old.
* Bad controlled mother's diabetes (at least two digits of blood glucose <180 mg/dl per day), bad alimentation control and/or non-adherence.

Ages: 6 Hours to 20 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time of cord separation | 15 days
  Examine the differences in the cord separation time between alcohol 70º and soap.

SECONDARY OUTCOMES:
Umbilical cord infection | 28 days
Omphalitis | 28 days
Pneumonia | 28 days
Diarrhea | 28 days
Tetanus | 28 days
Neonatal mortality | 60 days
Hospital admissions | 60 days
Emergency department admissions | 60 days
Unscheduled consultations | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Lara Perez, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain